CLINICAL TRIAL: NCT00405314
Title: Prehospital CPAP Versus Usual Care for Acute Respiratory Failure: a Randomized Controlled Trial
Brief Title: Prehospital CPAP vs. Usual Care for Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAL06-04
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Respiratory Insufficiency; Hypoxia
Keywords: respiratory failure; non invasive ventilation; prehospital; endotracheal intubation; continuous positive airway pressure
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

INTERVENTIONS:
Device: Continuous positive airway pressure ventilation mask

SUMMARY:
The purpose of this study is to evaluate the effectiveness of continuous positive airway pressure ventilation when applied by paramedics to individuals with severe breathing difficulties in the prehospital setting.

DETAILED DESCRIPTION:
Continuous positive airway pressure ventilation (CPAP) has been shown to be effective in avoiding endotracheal intubation (ETI) for patients with acute respiratory failure in hospital but despite several case series, the effectiveness of the prehospital application of CPAP by paramedics has not been studied in a randomized fashion. We performed a prospective, randomized, non blinded trial to determine whether patients in acute respiratory failure treated with CPAP in the prehospital setting had lower overall ETI rates than those treated with standard care.

ELIGIBILITY:
Inclusion Criteria:

* severe dyspnea
* respiratory rate >25 breaths/minute
* hemodynamically stable
* able to cooperate with ventilatory support measures
* assessed by paramedics as being in urgent need of ETI and/or manual positive pressure ventilation
* a trip destination of the QEII Health Sciences Center or Dartmouth General Hospital

Exclusion Criteria:

* require ETI for immediate airway protection
* respiratory rate < 8 breaths/minute
* evidence of hemodynamic instability
* cardiac ischemia
* any chest pain within 3 hours of presentation
* valid "do not resuscitate" advanced directive
* an inadequate supply of portable oxygen

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2002-07; Study Completion 2006-03

PRIMARY OUTCOMES:
proportion of patients in each group endotracheally intubated prior to hospital discharge or death

SECONDARY OUTCOMES:
mortality
critical care unit length of stay
hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: James Thompson, MD, Principal Investigator — University of British Columbia
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Wang HE, Yealy DM. Out-of-hospital endotracheal intubation: where are we? Ann Emerg Med. 2006 Jun;47(6):532-41. doi: 10.1016/j.annemergmed.2006.01.016. Epub 2006 Feb 28. PMID 16713780
- [Background] Winck JC, Azevedo LF, Costa-Pereira A, Antonelli M, Wyatt JC. Efficacy and safety of non-invasive ventilation in the treatment of acute cardiogenic pulmonary edema--a systematic review and meta-analysis. Crit Care. 2006;10(2):R69. doi: 10.1186/cc4905. PMID 16646987
- [Background] Hubble MW, Richards ME, Jarvis R, Millikan T, Young D. Effectiveness of prehospital continuous positive airway pressure in the management of acute pulmonary edema. Prehosp Emerg Care. 2006 Oct-Dec;10(4):430-9. doi: 10.1080/10903120600884848. PMID 16997770
- [Derived] Thompson J, Petrie DA, Ackroyd-Stolarz S, Bardua DJ. Out-of-hospital continuous positive airway pressure ventilation versus usual care in acute respiratory failure: a randomized controlled trial. Ann Emerg Med. 2008 Sep;52(3):232-41, 241.e1. doi: 10.1016/j.annemergmed.2008.01.006. Epub 2008 Apr 3. PMID 18387700